CLINICAL TRIAL: NCT02427867
Title: Ischaemic PReconditioning In Non Cardiac surgEry
Acronym: PRINCE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Associate Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRINCE/43/OSR
Record Dates: First submitted 2015-04-15; First posted 2015-04-28 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Ischemia; Surgery
Keywords: remote ischemic preconditioning; non cardiac surgery; myocardial ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- remote ischemic preconditioning (Experimental): Three cycles of 5 minutes ischemia will be applied to the upper left arm (or right arm or legs if the left arm will not be deemed suitable by the attending physician), achieved by inflation of a blood-pressure cuff to 200 mm Hg, followed by 5 minutes reperfusion while the cuff will be deflated.
  Interventions: Other: Remote ischemic preconditioning
- no ischemic preconditioning (Placebo Comparator): The cuff will be placed around the arm but not inflated.
  Interventions: Other: no ischemic preconditioning

INTERVENTIONS:
Other: Remote ischemic preconditioning
  Arms: remote ischemic preconditioning
Other: no ischemic preconditioning
  Arms: no ischemic preconditioning

SUMMARY:
Several randomized trials suggested a cardioprotective beneficial effect (eg reduction in cardiac troponin release) of remote ischemic preconditioning in cardiac surgery.

Remote ischemic preconditioning by brief episodes of ischemia and reperfusion in a remote organ or vascular territory provides protection from injury by myocardial ischemia and reperfusion. In the translation of remote ischemic preconditioning from bench to bedside, the first proof of principle and small randomized controlled trials have shown a decreased release of myocardial biomarkers after aortic, congenital cardiac, adult valve and coronary artery by-pass graft surgery. This reduction in cardiac biomarkers release translated into better survival in a recent randomized trial performed in cardiac surgery. No clinical trial on remote ischemic preconditioning in non-cardiac surgery setting has been performed so far.

The investigators study wants to test, for the first time, the hypothesis that remote ischaemic preconditioning is effective in reducing cardiac damage in high risk patients undergoing non-cardiac surgery. Remote ischaemic preconditioning will be achieved by inflation of a blood-pressure cuff to 200 mm Hg to the upper arm for 5 minutes, followed by 5 minutes reperfusion while the cuff will be deflated. General anesthesia will be induced and maintained without using propofol in both groups. Cardiac troponin will be used as marker of cardiac damage. If the results of a reduction in postoperative cardiac troponin release and perioperative cardiac ischaemic events will be confirmed in a non-cardiac surgery setting, the investigators could improve a strategy to prevent perioperative cardiac complication easy to apply, safe and low cost.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* intermedial and high risk non cardiac surgery
* general anesthesia
* ongoing or recently suspended antiplatelet therapy

Exclusion Criteria:

* pregnancy
* planned locoregional anesthesia without general anesthesia
* unstable or ongoing angina
* recent (< 1 month) or ongoing acute myocardial infarction
* inclusion in other randomised controlled studies in the previous 30 days
* peripheral vascular disease affecting the upper limbs
* cardiac surgery

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1217 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2025-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
cardiac troponin | Hospital - approximately 1 week
  elevation of cardiac troponin after non-cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Zangrillo, Prof., Study Chair — Vita-Salute University of Milan
Locations (26):
- Xijing Hospital, Xi'an, China
- Fundación Cardioinfantil-Instituto de Cardiología, Bogotá, Colombia
- University Hospital Centre Zagreb, Zagreb, Croatia
- Italy (14):
  - Humanitas Clinical Institute, Rozzano, Lombardy
  - Valle Olona Po hospital, Busto Arsizio, Varese
  - Ospedale Cardinal Massaia, Asti
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - E.O. Ospedali Galliera, Genova
  - IRCCS San Raffaele Scientific Institute, Milan
  - Fondazione IRCCS. Istituto Neurologico Carlo Besta, Milan
  - Università degli studi della Campania Luigi Vanvitelli, Napoli
  - Azienda Universitaria Ospedaliero Pisana, Pisa
  - A.O.U. Pisana, Pisa
  - Fondazione Policlinico Universitario Campus Bio-Medico di Roma, Rome
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - ULSS 4 Veneto Orientale, Ospedale di San Donà di Piave, San Donà di Piave
  - Azienda Sanitaria Universitaria Friuli Centrale "Santa Maria della Misericordia", Udine
- Astana Medical University, Astana, Kazakhstan
- Russia (5):
  - Loginov Moscow Clinical Scientific Center, Moscow
  - Oncological Center No. 1 of the S. S. Yudin City Clinical Hospital of the Moscow Department of Health, Moscow
  - I.M. Sechenov First Moscow State Medical, Moscow
  - V.Negovsky Reanimatolgy Research Institute, Moscow
  - Saint-Petersburg State University Hospital, Saint Petersburg
- Institute of Cardiovascular Diseases "Dedinje", Belgrade, Serbia
- National University Hospital, Singapore, Singapore
- Ospedale Regionale di Lugano, Lugano, Switzerland

REFERENCES:
- [Background] Massimiliano Greco, Gaetano Lombardi, Aidos Konkayev, Claudia Brusasco, Chong Lei, Agostino Roasio, Nerlep Rana, Hugo A. Mantilla-gutierrez, Marco Micali, Gordana Gazivoda, Michela Gandini, Lian Kah Ti, Stefano Bosso, Maiya Konkayeva, Francesco Meroi, Lini Wang, Andrea Russo, Sergey Efremov, Giuseppe Fresta, Levan Berikashvili, Francesca Livi, Ivan Šitum, Fabio Guarracino, Elizaveta Leonova, Francesca Cavenago, Maria Shemetova, Edoardo Cristallo, Anastasia Smirnova, Lorenzo Schiavoni, Valerii Subbotin, Nicoletta Boffa, Giuseppe Giardina, Michele Introna, Cristina Nakhnoukh, Remo Daniel Covello, Marina Pieri, Stefano Turi, Valentina Ajello, Fabrizio Monaco, Francesco Corradi, Andrey Yavorovskiy, Valery Likhvantsev, Federico Longhini, Tiziana Bove, Rinaldo Bellomo, Giovanni Landoni, Alberto Zangrillo, Rosalba Lembo. Remote ischemic preconditioning in non-cardiac surgery (PRINCE): a multinational, double blind, sham-controlled, randomized clinical trial. Signa Vitae. 2024. 20(12);1-9. https://www.signavitae.com/articles/10.22514/sv.2024.151
- [Derived] Greco M, Lombardi G, Brusasco C, Pieri M, Roasio A, Monaco F, Berikashvili L, Belletti A, Meroi F, Fresilli S, Kabibulatov A, Giardina G, Russo A, Oliva FM, Efremov S, Lembo R, Wang L, Vietri S, Momesso E, D'Amico F, Kadantseva K, Labanca R, Ryzhkov P, Marmiere M, Subbotin V, Pruna A, Rana N, Livi F, Mantilla-Gutierrez H, Guarracino F, Schiavoni L, Situm I, Micali M, Bosso S, Smirnova A, Fresta G, Cherednichenko A, Beretta L, Monti G, Ti LK, Sansone P, Corradi F, Cecconi M, Yavorovskiy A, Lei C, Konkayev A, Bove T, Likhvantsev V, Zangrillo A, Landoni G, Bellomo R, Covello RD, Turi S; PRINCE Study Group. Effect of Remote Ischemic Preconditioning on Myocardial Injury in Noncardiac Surgery: The PRINCE Randomized Clinical Trial. Circulation. 2025 Oct 28;152(17):1194-1205. doi: 10.1161/CIRCULATIONAHA.125.075254. Epub 2025 Jun 13. PMID 40511609
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250